CLINICAL TRIAL: NCT02753192
Title: Dysarthria in Parkinson's Disease: Lusophony vs. Francophony Comparison
Acronym: FraLusoPark
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre National de la Recherche Scientifique, France (Other)
Collaborators: Instituto de Medicina Molecular João Lobo Antunes (Other)
Responsible Party: Principal Investigator, Serge Pinto, Dr. Serge Pinto, Ph.D., Centre National de la Recherche Scientifique, France
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 13017; ANR-13-ISH2-0001-01 (Other Grant/Funding Number: ANR); FCT-ANR/NEU-SCC/0005/2013 (Other Grant/Funding Number: FCT)
Record Dates: First submitted 2016-04-25; First posted 2016-04-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Parkinson's Disease; Dysarthria; Speech; Cross-language; Medical Treatment; Disease Progression
MeSH Terms: conditions — Parkinson Disease; Dysarthria; Speech; Disease Progression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients (Other): Individuals with PD will be enrolled in the study in Aix-en-Provence, France (N = 60) and Lisbon, Portugal (N = 60). Their global motor disability and orofacial motor functions will be assessed with specific clinical rating scales, without (OFF) and with (ON) medical treatment. Two groups of 60 healthy age-matched volunteers will provide the reference for between-group comparisons.
  Interventions: Other: Patients

INTERVENTIONS:
Other: Patients — Individuals with PD will be enrolled in the study in Aix-en-Provence, France (N = 60) and Lisbon, Portugal (N = 60). Their global motor disability and orofacial motor functions will be assessed with specific clinical rating scales, without (OFF) and with (ON) medical treatment. Two groups of 60 healthy age-matched volunteers will provide the reference for between-group comparisons. Along with the clinical examinations, several speech tasks will be recorded to obtain acoustic and perceptual measures. Self-evaluation questionnaires will be used to assess the psychosocial impact of dysarthria on quality of life.

SUMMARY:
Parkinson's disease (PD) affects between 1% and 2% of the world's population aged 60 and older; in Europe the prevalence is around 150 PD patients per 100,000 individuals. PD is classically characterized by a symptomatic triad that includes rest tremor, akinesia and hypertonia and although the motor expression of the symptoms involves mainly the limbs, the muscles implicated in speech production are also subject to specific dysfunctions. Motor speech disorders, so-called dysarthria, can thus be developed by PD patients. The main objective of our project is to evaluate the physiological parameters (acoustics), perceptual markers (intelligibility) and psychosocial impact of dysarthric speech in PD, in the context of language (French vs. Portuguese) modulations. Acoustic parameters are expected to be physiologically-based, linked with the motoric aspects of dysarthric speech. The same degree of impairment of such parameters should be associated with the pathology and be present universally in all patients, even if they speak different languages; that should be also the case of prosodic markers, whereas impairment of speech intelligibility may participate to the psychosocial impact in communication alteration.

PD patients will be enrolled in the study in Aix-en-Provence (N = 60) and Lisbon (N = 60). Their global motor disability will be assessed with dedicated clinical rating scales, without (off) and with (on) pharmacological treatment. Two groups of 60 healthy age-matched volunteers will provide the normal reference for between-group comparisons. Along with the off and on medication clinical examinations, several speech tasks will be recorded. Moreover, speech organ functions will also be assessed during the same examination. The psychosocial impact of dysarthria will be evaluated via self-questionnaires; it will be analysed a posteriori, as well as the speech intelligibility evaluation, and both will strengthen the overall speech assessments. This global investigation will represent a unique opportunity to provide the most precise and reliable description of PD patients' speech and its impacts on intelligibility and quality of life. Challenging and interdisciplinary aspects are combined in our project, which original cross-linguistic approach involves an international collaboration definitely new in the field of motor speech disorders.

DETAILED DESCRIPTION:
Background - Individuals with Parkinson's disease (PD) have to deal with several aspects that contribute to voice and speech decline and thus, alteration of communication ability during the course of the disease: (i) The orofacial motor dysfunction, so-called dysarthria, which depends on the neurodegenerative processes; (ii) The effects of the medical treatment, which vary according to the disease stage; and (iii) The particular speech modifications that can be language-specific, i.e. dependent on the language spoken by the patients. The main objective of the FralusoPark project is to evaluate changes in dysarthric speech in PD as a result of medical treatment and disease duration using acoustic parameters (voice and prosody), perceptual markers (intelligibility), and patient-based outcomes (the psychosocial impact on quality of life) in two different languages (French vs. European Portuguese).

Methods - Individuals with PD will be enrolled in the study in Aix-en-Provence, France (N = 60) and Lisbon, Portugal (N = 60). Their global motor disability and orofacial motor functions will be assessed with specific clinical rating scales, without (OFF) and with (ON) medical treatment. Two groups of 60 healthy age-matched volunteers will provide the reference for between-group comparisons. Along with the clinical examinations, several speech tasks will be recorded to obtain acoustic and perceptual measures. Self-evaluation questionnaires will be used to assess the psychosocial impact of dysarthria on quality of life.

Discussion - Our three a priori hypotheses are the following: (i) Global acoustic features are altered similarly in French and Portuguese individuals with PD; (ii) Language-specific prosodic patterns might be altered differently according to the language spoken by the patients; and (iii) The impact of speech disorders on intelligibility and quality of life depends on the cultural and linguistic environment. The study combines an interdisciplinary and cross-linguistic approach to study motor speech disorders and will allow for a better understanding of the progression of speech symptoms in PD and their response to medical treatment. It will provide recommendations on how to assess speech and voice disorders in individuals with PD in order to monitor symptom progression and management.

ELIGIBILITY:
Inclusion Criteria:

All participants

* Age between 35 and 85 years old
* Good cooperation
* Ability to understand the information sheet
* Given signed consent
* Affiliation to a medical-social insurance regimen
* Other stable medical problems not interfering with the proposed study

Only for patients:

* Absence of any neurological, psychiatric or behavioral pathology
* Idiopathic Parkinson's disease
* Absence of medication-induced psychosis, severe depression or dementia

Exclusion Criteria:

All participants

* Illiteracy
* French/Portuguese not as native language, or bilingual participants
* Participant under tutorship or guardianship, or any other administrative or legal measure
* No cooperation or withdrawn consent
* Cognitive deficits, depression, psychosis or behavioral, neurological, medical, psychological disorders that may interfere with vital prognostic and evaluations

Only for patients:

* Non-idiopathic Parkinson's disease
* (Too) severe motor impairment impeding to participate in the study

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Global acoustic features | Day of assessment
  Participants are recorded while performing several tasks and the acoustic measures characterize dimensions of aero-phonatory control. For example, for the steady vowel /a/ phonation, two kinds of measures will be extracted: First, for a macro-analysis: fundamental frequency (F0, Hertz) and F0 variation (%); and second, for a micro-analysis: perturbation measures such as jitter factor (%), absolute shimmer (dB), and harmonics-to-noise ratio (HNR, %). For the maximal phonation time, the longest duration (in seconds) of the sustained vowel /a/ will be extracted.
Clinical features | Day of assessment
  The neurological assessment is the Unified Parkinson's Disease Rating Scale, using the revised version provided by the Movement Disorders Society (MDS-UPDRS). The FDA2 is used to assess the functions of the speech organs, reflecting the state of the muscular effectors involved in speech production.
Patient-reported outcome measures | Day of assessment
  Patient-reported outcome measures (PROMs), such as the Dysarthria Impact Profile (DIP), are used to obtain self-reported information about the functional impact of their speech/communication impairment. Additional self-assessments focus on the patients' perception of their quality of life (the 39-Item Parkinson's Disease Questionnaire [PDQ-39]) and on how voice/speech impairment may induce a handicap (Voice Handicap Index, VHI). The French and European Portuguese adapted DIP, VHI and PDQ-39 will be used in our study. The Patient Global Impression (PGI) scoring, and the Beck Depression Inventory (BDI) are also administered. The MDS-UPDRS also includes a patient self-assessment (sections 1.B and 2), which are administered together with the other questionnaires under medication.

SECONDARY OUTCOMES:
Prosodic analyses | Day of assessment
  Specific analyses of language-induced prosodic variations.
Intelligibility of speech | Day of assessment
  Refined intelligibility evaluation using an auditory jury.

CONTACTS AND LOCATIONS:
Overall Officials: Serge Pinto, Ph.D., Principal Investigator — Laboratoire Parole et Langage, Aix-en-Provence, France; Joaquim J Ferreira, M.D, Ph.D., Principal Investigator — Instituto de Medicina Molecular, Lisobon School of Medicine, Lisbon, Portugal
Locations (3):
- Centre Hospitalier du Pays d'Aix - Service de Neurologie, Aix-en-Provence, France
- Portugal (2):
  - Santa Maria University Hospital, Lisbon
  - Campu Neurologico Senior (CNS), Torres Vedras

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Derived] Pinto S, Cardoso R, Sadat J, Guimaraes I, Mercier C, Santos H, Atkinson-Clement C, Carvalho J, Welby P, Oliveira P, D'Imperio M, Frota S, Letanneux A, Vigario M, Cruz M, Martins IP, Viallet F, Ferreira JJ. Dysarthria in individuals with Parkinson's disease: a protocol for a binational, cross-sectional, case-controlled study in French and European Portuguese (FraLusoPark). BMJ Open. 2016 Nov 17;6(11):e012885. doi: 10.1136/bmjopen-2016-012885. PMID 27856480